CLINICAL TRIAL: NCT03846635
Title: Handheld Infrared Thermometer to Evaluate Cellulitis
Acronym: HI-TEC
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Todd Lee, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2019-4850
Record Dates: First submitted 2019-02-08; First posted 2019-02-19 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Cellulitis; Cellulitis of Arm; Cellulitis of Leg
Keywords: Cellulitis; Temperature; Venous Stasis; Lymphedema
MeSH Terms: conditions — Cellulitis; Varicose Ulcer; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Suspected Cellulitis: Patients who undergo an infectious diseases consultation for suspected cellulitis of the upper or lower limbs are eligible to be enrolled. Patients who consent to participation will have chart data extracted and undergo a skin surface temperature measurement of the affected area and surrounding skin using a commercially available infrared thermometer. The dimensions of suspected cellulitis are also measured.
  Patients with cellulitis admitted to hospital undergo daily measurements of temperature and dimensions. These patients are also asked standardized questions about their symptoms based on the patient global impression of improvement scale.

SUMMARY:
It can be difficult to differentiate cellulitis from non-infectious mimics, like venous stasis. One way of determining the difference is feeling skin surface temperature. However, this is a subjective measure that is inherently unreliable. It might be possible to objectify this measurement by using a non-contact infrared thermometer at the bedside.

The goal of this study is therefore to assess whether objective difference in skin surface temperature in an area of suspected cellulitis, relative to non-affected skin, has diagnostic utility. It will use the diagnosis of cellulitis by an infectious diseases physician as the gold standard and compare blinded temperature difference between affected and unaffected limbs to that standard. It is hypothesized that measurement of skin surface temperature by non-contact infrared thermometer will help differentiate cellulitis from many non-infectious conditions that mimic cellulitis.

For patients who are hospitalized, the study also plans to see whether a change in this temperature difference is predictive of response to treatment when compared to the FDA standard for early response and patient reported symptoms.

This is a pragmatic, prospective cohort study. Patients with suspected cellulitis who receive an infectious diseases consult (in the emergency room or urgent clinic) will be approached for consent and enrollment. The goal is to enroll approximately 50 patients with a minimum of 10-15 cases of non-cellulitis.

These measurements will not be made available to the treating teams. This is an observational study only comparing the potential value of these measurements to usual clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* English or French-speaking;
* Received an infectious diseases consultation to evaluate proven or suspected cellulitis of the upper or lower extremity, either unilaterally or bilaterally;
* Either no empiric antimicrobials received or, at most, antimicrobials begun within 24 hours of notification for enrollment.

Exclusion Criteria:

* Presumptive diagnosis of a soft tissue infection of the trunk, head or neck that does not also involve a limb;
* Patients with only one limb;
* Patients with significant neuropathies or autonomic syndromes that might affect thermoregulation, such as severe diabetic neuropathy or diabetic dysautonomia, neurologic neoplasms and known vitamin deficiencies;
* Soft tissue infections requiring definitive surgical source control, such as abscesses or necrotizing fasciitis.

  * Septic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As above, our patient population includes patients aged 18 years and older who can communicate in English or French who receive an infectious diseases consultation for cellulitis of a limb.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Difference in skin temperature between affected and contra-lateral limb | Skin temperature measurement at time of enrolment
  The difference in skin surface temperature measured at the site of suspected cellulitis versus the same location on the contra-lateral limb will be compared to the treating physician's diagnosis of cellulitis/not cellulitis.

SECONDARY OUTCOMES:
Change in Skin Temperature | Serial measurements daily until (a) discharge or (b) cure of cellulitis whichever comes first up to a maximum of 14 days
  For patients who are hospitalized for antibiotic therapy, skin surface temperature of the affected area will be measured on a daily basis.
Change in Maximal Dimensions of Cellulitis | Serial measurements daily until (a) discharge or (b) cure of cellulitis whichever comes first up to a maximum of 14 days
  For patients who are hospitalized for antibiotic therapy, cellulitis length and width dimensions (FDA early response criteria for cellulitis) will be measured on a daily basis.
Clinical symptoms of cellulitis as measured by the patient global impression of change scale | Serial evaluations daily until (a) discharge or (b) cure of cellulitis whichever comes first up to a maximum of 14 days
  Patient global impression of change scale (PGIC) as compared to their initial presentation. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD MPH FACP, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03846635/SAP_001.pdf
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03846635/Prot_002.pdf